CLINICAL TRIAL: NCT00369499
Title: STOP PAIN: Septal Closure of PFO - Does it Prevent Migraine?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients/ ethical concerns
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV05003PC
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

INTERVENTIONS:
Device: PFO Closure

SUMMARY:
The primary objective of this Study is to compare the effect of transcatheter device closure of atrial shunting to a non-closure control group over a period from cessation of procedure related medication at 3 months until 9 months post randomization by determining the proportion of patients that experience a 50% or more reduction in the baseline monthly migraine attack frequency in each group.

ELIGIBILITY:
Inclusion Criteria:

* Migraine history of at least 1 year.
* Migraine patients experiencing at least 2 migraine attacks per month.
* Migraine patients experiencing at least 1 migraine attack with aura per month.
* Failure of or intolerance to at least 2 classes of prophylactic migraine medication evaluated in adequate, approved medication trials. At least one of the classes shall come from beta-blockers, anticonvulsants, calcium channel blockers and tricyclic antidepressants.
* Aged 18 - 50 years and of legal age in the host country.
* The patient or legal guardian has signed a study specific informed consent form agreeing to data collection and follow-up requirements.
* The patient agrees to abstain from starting prophylactic migraine medication or agrees to maintain existing prophylactic migraine medication without changing dose or drug from entering the baseline period throughout the duration of the study until final assessments.
* Documented right to left shunt that is suitable for device closure.

Exclusion Criteria:

* Taking migraine preventative medication for conditions other than migraine.
* History of 15 or more headache days per month.
* 8 or more non-migraine headache days per month.
* Overuse of acute headache medication (use on 10 or more days per month).
* Patient has severe central nervous system disease such as seizure disorder, inflammatory disease of the central nervous system, or a previous stroke.
* Previous surgical or device closure of a PFO or ASD.
* Artificial heart valve.
* Pacemaker or ICD implanted within past 3 months.
* Anatomic variant that could affect successful deployment such as coronary sinus, pulmonary veins, Chiari network.
* Uncontrolled bacteremias or dental or surgical procedure within past 30 days or planned within study period.
* Allergy to contrast media, and/or to any component of the device to be used.
* Contraindicated for any medication used during or after the procedure.
* History of atrial fibrillation or atrial flutter (chronic or paroxysmal).
* Patient is enrolled or intends to participate in another clinical study (of an investigational drug or device, new indication for an approved drug or device, or requirement of additional testing beyond standard clinical practice) during the study or within four weeks prior to his/her enrollment in the study.
* Patient is undergoing dialysis for renal failure.
* Patient has NYHA class 3 or 4 cardiac failure.
* Patient is pregnant, or intends to become pregnant during the trial period.
* Patient requires anticoagulation therapy for a concomitant condition.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 656 (Estimated)
Dates: Start 2007-03; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Mean values of the number of monthly migraine periods, with or without aura.

SECONDARY OUTCOMES:
Mean values of monthly migraine frequency with or without aura.
Quality of life using a Headache Impact Test Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ferrari, Prof., Principal Investigator — Leiden University Medical Centre; Horst Sievert, Prof., Principal Investigator — CardioVascular Center Frankfurt, Sankt Katharinen
Locations (1):
- CardioVascular Center Frankfurt, Sankt Katharinen, Frankfurt, Germany